CLINICAL TRIAL: NCT05014984
Title: WOOP VA: Mental Contrasting With Implementation Intentions to Promote Weight Management in Primary Care
Brief Title: WOOP VA: Promoting Weight Management in Primary Care
Acronym: WOOP VA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIR 20-153
Record Dates: First submitted 2021-08-04; First posted 2021-08-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: obesity; primary care; Weight management
MeSH Terms: conditions — Obesity | interventions — Exercise; Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study staff, investigators, and outcome assessors will be blinded to the intervention arm. The lay health coach interventionist and the participant will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telephone Delivered MOVE!/TeleMOVE! (Active Comparator): During the baseline visit, Veterans randomized to the control arm will receive only the standard information about MOVE!/TeleMOVE!, diet, and physical activity delivered by the same lay educators. They will not learn the WOOP technique as detailed below. Data collection during study visits will be at the same timepoints in both arms.
  Interventions: Behavioral: telephone-delivered, telehealth-delivered, and or in-person MOVE! or TeleMOVE!; Behavioral: Information About Diet, Physical Activity, and Weight Management (Baseline Visit - 10 minutes): All
- Mental Contrasting with Implementation Intentions (WOOP) plus MOVE! /TeleMOVE! (Experimental): At the baseline visit, a lay educator will teach the WOOP technique in-person using protocols adapted from our prior work. After, to support WOOP practice, the lay educator will schedule and provide 3 follow-up telephone check-ins with the Veteran. This arm will also receive telephone-delivered MOVE!/TeleMOVE!
  Interventions: Behavioral: mental contrasting with implementation intentions; Behavioral: telephone-delivered, telehealth-delivered, and or in-person MOVE! or TeleMOVE!; Behavioral: Information About Diet, Physical Activity, and Weight Management (Baseline Visit - 10 minutes): All; Behavioral: Telephone MCII Check-ins (30 minutes at 3 days, 4 weeks, and 2 months after baseline visit)

INTERVENTIONS:
Behavioral: mental contrasting with implementation intentions — To deliver MCII, Dr. Oettingen developed a step-wise procedure called WOOP (Wish, Outcome, Obstacle, Plan; Figure 1). In a quiet setting, patients identify an important wish (e.g., losing weight) and then name and vividly imagine the best outcome (e.g., feeling healthier). Next, they name a current internal obstacle (e.g., urge to eat when feeling stressed) and try to vividly imagine their experience when they encounter this obstacle. Finally, they address their obstacle with an if-then plan specifying when, where, and how to overcome it (e.g., "If I have the urge to eat when feeling stressed, I will go for a walk)" and then imagine themselves experiencing the obstacle and carrying out the action of surmounting it. To facilitate use of the WOOP technique, Dr. Oettingen developed a free, publicly available WOOP app
  Other Names: WOOP (Wish, Outcome, Obstacle, Plan)
  Arms: Mental Contrasting with Implementation Intentions (WOOP) plus MOVE! /TeleMOVE!
Behavioral: telephone-delivered, telehealth-delivered, and or in-person MOVE! or TeleMOVE! — MOVE! is a national VA weight management and health promotion program to improve the quality of life of Veterans.6,75 This effective program encourages healthy eating behavior and increased physical activity. MOVE! will be delivered via telephone (16 sessions) by existing staff consistent with national MOVE! program guidelines. The program has 16 modules and will offered weekly, but Veterans will be able to make up sessions at their own pace if they miss one. MOVE! staff use the MOVE! facilitator guide that provides instruction on delivering the program via telephone. Update as of 11-2023, the New York Harbor VA paused their offering of telephone-delivered MOVE!. Participants in both arms are offered the in-person or video-delivered MOVE! program. For participants who do not want or are unable to attend group-based MOVE!, they are offered TeleMOVE!.
Behavioral: Information About Diet, Physical Activity, and Weight Management (Baseline Visit - 10 minutes): All — All participants will receive handouts that they review with a lay educator on weight management, adapted from the educational materials developed for our FIReWoRk Study. Topics include losing weight at a healthy rate, setting a 6-month weight loss goal of 5-10%, limiting sugar-sweetened beverages and portion sizes, making better choices when eating at restaurants, self-monitoring diet and weight, and participating in at least moderate-intensity physical activities.
Behavioral: Telephone MCII Check-ins (30 minutes at 3 days, 4 weeks, and 2 months after baseline visit) — The lay educator will review and practice the WOOP technique based on protocols from prior studies. To probe Veterans' comprehension, the lay educator will ask for their four steps and ask about their WOOP use and experiences. If needed, the lay educator will help the Veteran to create a new WOOP for the next month and address any questions and concerns about using WOOP.
  Arms: Mental Contrasting with Implementation Intentions (WOOP) plus MOVE! /TeleMOVE!

SUMMARY:
Approximately 40% of Veterans have obesity and are at increased risk for cardiometabolic disease. Intensive lifestyle-based weight management programs can lead to clinically significant ( 5%) weight loss. The VA's MOVE! program is effective for promoting weight loss and behavior change for those who attend. Unfortunately, MOVE! has low enrollment and high attrition due to several obstacles including low motivation. Mental Contrasting with Implementation Intentions (MCII) is an innovative strategy developed over 20 years of research that uses imagery to increase motivation for behavior change. MCII can be implemented in primary care settings using an easy to teach technique called "WOOP" (Wish, Outcome, Obstacle, Plan) that Veterans then use regularly on their own with the help of paper-based tools or the WOOP app. The research team will evaluate the efficacy and implementation of MCII when combined with telephone-delivered MOVE! vs. telephone-delivered MOVE! alone to enhance weight management outcomes for Veterans in primary care.

DETAILED DESCRIPTION:
Background: Approximately 40% of Veterans have obesity. Intensive weight management programs such as MOVE! promote clinically significant weight loss, but only 3-7% of eligible Veterans attend. Low enrollment and high attrition are due to obstacles such as travel, cost, and motivation. Developed through over 20 years of research, Mental Contrasting with Implementation Intentions (MCII) is a novel, evidence-based intervention to increase motivation and behavior change. MCII has been shown to increase physical activity and consumption of fruits and vegetables and promote weight loss, and the research team recently demonstrated that MCII is feasible and acceptable to Veterans for weight management. However, has not been tested adequately within primary care nor demonstrated weight loss in Veterans. The investigators propose to evaluate the efficacy and implementation of MCII for behavior change and weight loss in Veterans within primary care when combined with the VA MOVE! Program.

Significance/Impact: This proposal aligns with the VA HSRD "primary care practice and management of complex chronic diseases" funding priority. Primary care providers and PACT members do not provide sufficient counseling to increase engagement with the MOVE! Program. MCII can be taught by lay educators and can be delivered in conjunction with MOVE! and other weight management treatments.

Innovation: MCII is innovative in its use of imagery, ease of delivery by lay educators, novel mechanisms of action (via non-conscious motivational and cognitive processes), and ability to be combined with other programs. Veterans can practice MCII on their own in under 10 minutes. MCII uses a standardized, 4-step imagery procedure called WOOP that can be taught in 30 minutes. Veterans can then continue to use WOOP regularly, with the assistance of a WOOP App and website containing video-, audio-, and paper-based tools. This study will be the first randomized controlled trial of MCII within primary care and the first RCT to test the efficacy and implementation of MCII for weight management when combined with MOVE! in Veterans.

Specific Aims: 1. Compare the impact of MCII + MOVE!/TeleMOVE! vs. MOVE!/TeleMOVE! alone on percent weight change and waist circumference at 6 and 12 months. 2. Compare the impact of MCII + MOVE!/TeleMOVE! vs. MOVE!/TeleMOVE! alone on MOVE!/TeleMOVE! program attendance, healthy eating, and physical activity at 6 and 12 months. 3. Evaluate implementation of MCII. The investigators will use the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework to evaluate implementation barriers, facilitators, and outcomes of MCII.

Methodology: The investigators will enroll 405 Veterans and randomize 366 Veterans at the patient level within primary care to either MCII + telephone-delivered MOVE!/TeleMOVE! (intervention) vs. telephone-delivered MOVE!/TeleMOVE! alone (control) at the Manhattan VA. At 6 and 12 months, participants will return to the clinic for a study visit where weight, diet, and physical activity will be assessed in both groups. The investigators will use intention-to-treat analyses.

Implementation/Next Steps: MCII is designed to be easily implemented in a variety of settings and for a variety of behaviors. Freely available online training materials will facilitate implementation. To guide future implementation and policy change, the research team will present data from Aim 3 implementation analyses and obtain input from Veteran stakeholders as well as local VA and NCP leaders. If found to be efficacious, the investigators will conduct hybrid effectiveness/implementation studies of MCII in a multi-site study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 (this age range represents MOVE!/TeleMOVE! eligibility);
* The most recent BMI of 30kg/m2 (with or without obesity-associated comorbidities) OR a BMI of 25kg/m2 with obesity-associated condition (heart diseases, hyperlipidemia, hypertension, cancer, diabetes, stroke, or osteoarthritis);
* at least 1 prior PCP visit in the past 24 months; access to a telephone; ability to travel to Manhattan VA for in-person evaluations at baseline, 6 and 12 months;
* desire to lose weight (Using 1-10 scale used in PI's other studies; minimum of 5/10);
* willingness to enroll in the MOVE!/TeleMOVE! program or any local/national VA program that support weight management.

Exclusion Criteria:

* Non-Veterans;
* a documented current history of active psychosis or other cognitive issues via ICD-10 codes;
* Diagnosed with Parkinson's disease and/or severe arthritis that might require joint or knee replacement in the next year;
* participating in a weight management study in the past year;
* taking an FDA-approved weight loss medication; Bupropion-naltrexone (Contrave) Liraglutide (Saxenda) Orlistat (Xenical)/alli Phentermine-topiramate (Qsymia) Phentermine Topiramate Lorcaserin / Belviq glucagon-like peptide 1 (GLP-1) agonists:

Diabetes drugs in the GLP-1 agonists class include:

Dulaglutide (Trulicity) Exenatide extended release (Bydureon) Exenatide (Byetta) Semaglutide (Ozempic) Semaglutide (Rybelsus) Liraglutide (Victoza) Lixisenatide (Adlyxin) Metformin to lose weight not for your diabetes;

* pregnancy;
* PCP stating that Veteran should not participate.
* Seeing a dietitian or MOVE!/TeleMOVE! Program attendance more than 3 times in the past year.
* Hospitalization within 90 days of enrollment.
* Anyone who is included in Dr. Jose Aleman weight management clinic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Weight Change | 6 months
  The research team will measure weight using a standardized protocol, taking the average of 2 weights in pounds, rounded to the nearest 0.1lb.

SECONDARY OUTCOMES:
Mean Percent Weight Change | 12 month
  The research team will measure weight using a standardized protocol, taking the average of 2 weights in pounds, rounded to the nearest 0.1lb.
Waist Circumference change | 6 and 12 months
  The RA will use an inelastic tape scaled in cm to measure the participant's waist circumference twice at the peak of the iliac crests, taking the average of the 2 measures rounded down to the nearest 0.25cm.
Healthy Eating Index change | baseline, 6 and 12 months
  The HEI-2015 is a diet quality index that measures alignment with the 2015-2020 Dietary Guidelines for Americans. To measure dietary intake at each time point, we will use an automated, cost-effective and valid 24-hour dietary recall instrument for measuring diet quality. The web-based Automated Self-Administered 24-Hour Recall (ASA24-2020), developed by the National Cancer Institute and first released in 2009 was modeled after the US Department of Agriculture's interviewer- administered Automated Multiple-Pass Method (AMPM). To limit participant burden, participants will perform one weekday measurement (self-administered in person with staff available to answer questions as needed) and one weekend measurement (self-administered at home). While at least three 24-hour recall measurements are considered the gold standard, two measurements are valid. If we cannot obtain a weekend measure, we will obtain two weekday measures and account for this in the analysis.
Physical Activity--Weekly minutes of Moderate to Vigorous Physical Activity (MVPA) | Baseline, 6 and 12 months
  The research team will use the ActiGraph Link (GT9X) accelerometer to objectively measure PA during a 7-day period. During an initial enrollment visit, RAs will place the Link monitor on the participant's non-dominant wrist and instruct the participant to measure PA for 24 hours a day for 7 days, except when swimming and bathing, and to return the monitor at the baseline visit two weeks later. We will use accelerometer data to report weekly minutes of MVPA.
MOVE! Attendance change | Baseline, 6 and 12 months
  A chart review will be done to verify the number of MOVE! sessions completed.
Change in Self Reported Physical Activity | Baseline, 6 and 12 months
  Self-reported weekly minutes of MVPA will be measured via the Global Physical Activity Questionnaire (GPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Melanie R. Jay, MD MS, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vandyousefi S, Oettingen G, Wittleder S, Moin T, Sweat V, Aguilar AD, Ruan A, Angelotti G, Wong L, Orstad SL, Illengberger N, Nicholson A, Lim S, Cansler R, Portelli D, Sherman S, Jay MR. Protocol for a prospective, randomized, controlled trial of Mental Contrasting with Implementation Intentions (MCII) to enhance the effectiveness of VA's MOVE! weight management program: WOOP (Wish, Outcome, Obstacle, Plan) VA. Contemp Clin Trials. 2024 Jun;141:107523. doi: 10.1016/j.cct.2024.107523. Epub 2024 Apr 10. PMID 38608752

DOCUMENTS (1):
  • Informed Consent Form (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05014984/ICF_000.pdf